CLINICAL TRIAL: NCT04143646
Title: New Technologies for Intensive Prevention Programs - NET-IPP
Acronym: NET-IPP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herzzentrum Bremen (Other)
Responsible Party: Principal Investigator, Dr. Harm Wienbergen, Head of the Bremen Institute for Heart and Circulation Research, Herzzentrum Bremen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIHKF 3
Record Dates: First submitted 2019-10-23; First posted 2019-10-29 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based prevention program (Active Comparator): Patients after myocardial infarction participate in a 12-months program with telemetric risk factor control, e-learning and E-Mail/App-contacts.
  In a substudy patients are further randomly assigned to disclosure of genetic risk vs. no disclosure.
  Interventions: Behavioral: Web-based prevention program
- Usual Care (No Intervention): Patients after myocardial infarction are treated following the standard of care (clinical practice as offered by general practitioners, cardiologists, etc.).

INTERVENTIONS:
Behavioral: Web-based prevention program — Telemetric control of risk factors, e-learning, contacts by e-mails/apps. If no response telephone calls.
  In a substudy evaluation of disclosure of genetic risk.
  Arms: Web-based prevention program

SUMMARY:
In a randomized trial patients hospitalized for myocardial infarction are prospectively enrolled and assigned to either a web-based intensive prevention program or usual care (1 : 1 randomization). The web-based program includes telemetric transmission of data on cardiocascular risk factors (physical activity, blood pressure, body weight) by patients to the study center, e-learning modules by the study center and repetitive electronic contacts by e-mails and apps between a prevention assistant and the patient.

In addition, genetic risk on cardiovascular events will be assessed in all patients of the intervention group by a polygenetic risk score (PRS). Patients of the intervention group are randomly assigned to disclosure of genetic risk vs. no disclosure. The study hypothesis is that disclosure of genetic risk improves cardiovascular risk factor control by increased patient motivation.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization due to acute myocardial infarction (ST-elevation or non-ST-elevation myocardial infarction) defined according to valid international guidelines
2. Access to internet and consent to participate in a web-based prevention program
3. Consent for genetic risk assessment for cardiovascular events and risk disclosure according to randomization

Exclusion Criteria:

1. Patient refusal or inability to give informed consent
2. Hemodynamically significant valvular heart disease
3. Exercise limitations due to clinical conditions not related to CAD (such as severe orthopedic disorders,..)
4. Any major non-cardiac condition that would adversely affect survival during the duration of the study (such as cancer with prognosis < 2 years,..)
5. Inability to cooperate with the protocol, including longterm follow-up
6. Chronic drug and alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of participants with serious adverse cardiovascular events | 24 months
  Serious adverse cardiovascular events are death (total and cardiovascular), resuscitations, strokes, myocardial infarctions, coronary revascularizations or hospitalizations due to unstable angina.

SECONDARY OUTCOMES:
LDL cholesterol | 24 months
  LDL cholesterol levels in mg per dl
Smoking status | 24 months
  Rate of participants who are active smokers in %
Physical inactivity | 24 months
  Caloric expenditure as assessed by IPAQ (International Physical Activity Questionnaire) in kilocalories per week
Blood pressure | 24 months
  Systolic and diastolic blood pressure measured in mmHg
Body mass index | 24 months
  Body mass index in kg/m² (calculated from body weight and height)
HbA1c | 24 months
  HbA1c levels in %

OTHER OUTCOMES:
Adherence to preventive medication | 24 months
  Rate of patients with lipid-lowering medication, antiplatelets (= aspirine, ticagrelor, prasugrel, clopidogrel)
Assessment of quality of life | 24 months
  Point score of the European Quality of Life 5 Dimensions (EQ5D) Questionnaire - Visual Analogue Scale (VAS). The Scale ranges from 0 to 100, with 100 indicating the best Quality of Life and 0 indicating the worst Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Herzzentrum Bremen, Bremen, Germany